CLINICAL TRIAL: NCT06192810
Title: Short- and Long-Term Outcomes of Adrenalectomy for Primary Aldosteronism in a Single UK Centre: Rear Mirror View
Brief Title: Short- and Long-term Outcomes of Adrenalectomy for Primary Aldosteronism
Status: Completed | Type: Observational
Sponsor: University College London Hospitals (Other)
Responsible Party: Principal Investigator, Alaa Abdelsalam, Principal investigator and clinical fellow, University College London Hospitals
Other Study IDs: 157714
Record Dates: First submitted 2023-11-14; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Primary Aldosteronism
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Procedure: Laparoscopic/open adrenalectomy

SUMMARY:
The proposed study is this. Short- and long-term outcomes of adrenalectomy for Primary Aldosteronism (PA) in a single centre. PA is a relatively common problem and considers as the commonest cause of secondary hypertension and can be successfully treated by adrenalectomy.

The investigators aim to gather clinical data routinely collected on participants with primary aldosteronism pre-operatively and post-operatively for a short and long term follow up.

DETAILED DESCRIPTION:
Retrospective analysis of data from a prospectively maintained database of participants with PA who underwent surgery between 1st January 1998 and 31st December 2022 at University College London Hospital, a tertiary referral centre for endocrinology and endocrine surgery.

The clinical pathway for screening, diagnosis and stratification for adrenalectomy varied through the 24 years and was based on concurrent recommendations, published evidence, changing local expertise and best practice at the time. Throughout this period diagnosis of PA in our centre was based on the presence of hypertension and hypokalaemia, high aldosterone level, suppressed renin activity and aldosterone and renin ratio (ARR) above 850. Currently a confirmatory test (for example, saline suppression test) recommended if the aldosterone is <550pmol/L but in the upper third of the normal range or the plasma renin is non-suppressed unless the patient presents with spontaneous hypokalaemia, plasma renin below detection levels and aldosterone concentration more than 550 pmol/L.

Stratification for adrenalectomy, once a diagnosis of PA was confirmed, included cross sectional imaging of adrenals with computed tomography (CT) or magnetic resonance imaging (MRI). Adrenal venous sampling (AVS) and/or later 11C Metomidate positron emission tomography-CT (PET-CT) scan was performed if imaging showed bilateral adrenal nodules. Surgery was recommended after discussion in the multidisciplinary team meeting (endocrinologist, endocrine surgeon, biochemists and radiologist).

During the very beginning of the study laparoscopic adrenalectomy was introduced and transperitoneal lateral technique was used to perform laparoscopic adrenalectomy using 3 ports on the left and 4 ports on the right side.

Participants included in the study were characterised preoperatively by their demographics (age, sex and ethnicity) clinical presentation (blood pressure), number of antihypertensive medications and biochemical tests (potassium, aldosterone, renin, ARR ratio).

Number and type of investigations (CT, MRI, AVS, Metomidate) used to stratify for surgery and the size of the adrenal nodules on cross sectional imaging was recorded. Process of stratification was presented as lateralisation to the left or right reached as a consensus between cross sectional imaging, AVS and nuclear medicine imaging.

Data on post operative surgical outcomes included conversion rate to open adrenalectomy, postoperative complications (Clavien-Dindo)and length of hospital stay.

Postoperative outcomes were assessed within 3 months of surgery (short term) and at least 60 months (long term). Data collected were blood pressure, number of antihypertensive medications, plasma concentration of potassium, aldosterone, renin and ARR ratio. Surgical outcomes were categorised using primary aldosteronism surgical outcome score (PASO) criteria of complete, partial or absent success for both clinical and biochemical cure which reflected remission, improvement or persistence of disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient underwent adrenalectomy as a management of primary aldosteronism
* Patient available for short term and long term follow up

Exclusion Criteria:

* medically treated patients
* not available for follow up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults diagnosed with primary aldosteronism and underwent surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 1998-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Short- and long-term assessment of clinical improvement in systolic and diastolic blood pressure | 3 months for short term and 5 years for long term
  Short- and long-term clinical changes for the following parameter:
  -Systolic and diastolic blood pressure measured in mmHg
Short- and long-term assessment of clinical improvement in number of antihypertensive medications in participants | 3 months for short term and 5 years for long term
  Short- and long-term clinical changes for the following parameter:
  -Number of antihypertensive medications

SECONDARY OUTCOMES:
Short- and long-term assessment of biochemical improvement in serum potassium level in participants | 3 months for short term and 5 years for long term
  Short-and long-term changes in biochemical parameter:
  -Serum Potassium level measured in mmol/L
Short- and long-term assessment of biochemical improvement in serum Aldosterone level in participants | 3 months for short term and 5 years for long term
  Short-and long-term changes in biochemical parameter:
  -Serum Aldosterone level measured in pmol/L
Short- and long-term assessment of biochemical improvement in serum Renin level in participants | 3 months for short term and 5 years for long term
  Short-and long-term changes in biochemical parameter:
  -Serum Renin level measured in nmol/L
Short- and long-term assessment of biochemical improvement in serum Aldosterone/Renin ratio (ARR) (pmol/nmol/L) level in participants | 3 months for short term and 5 years for long term
  Short-and long-term changes in biochemical parameters:
  -Serum Aldosterone/Renin ratio ARR (pmol/nmol/L)

IPD SHARING:
Plan to Share IPD: No